CLINICAL TRIAL: NCT04041180
Title: Incentive Spirometry and Pain in the Decompensation of Sickle Cell Disease: Impact on the Length of Stay. Prospective Observational Study
Brief Title: Impact on the Length of Stay in Incentive Spirometry and Pain in the Decompensation of Sickle Cell Disease: .
Acronym: SPIDO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2018-04
Record Dates: First submitted 2019-02-04; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Sickle Cell Disease; Pediatric
Keywords: Sickle cell disease; incentive spirometry; pain; children
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective observational study among sickle cell children aged 7 to 17 years, who face many experience of pain, pain will be assessed during incentive spirometry sessions. Then a relation between, inspiratory volume, pain and the length of hospital stay will be identified .

Currently, there is no scientific data regarding the correlation between acute pain during vaso-occlusive crisis, incentive spirometry and the impact on length of hospital stay. In fact, physiotherapist experience's in the pediatric department suggests that the pain expressed by the child is not always correlated with inspiratory capacity.

The absence of pain is one of the reasons for hospital discharge after decompensation in patients with sickle cell disease. However, no scientific study has linked incentive spirometry, pain and length of hospital stay.

Investigator assume that these children underestimate the real pain and its impact on breathing pattern, and presume that the maximal inspiratory volume during spirometry sessions will be a better reflect of pain than standard pain scale.

The aim of this study is to show that inspiratory volume would be a better indicator of discharge from hospitalization than actual pain scales.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell children aged 7 to 17 admitted to the pediatric ward
* Children receiving respiratory physiotherapy sessions under medical prescription
* Children hospitalized for more than 24 hours at the CHRO and benefiting from more than one physiotherapy session.
* Absence of opposition of one of the parents to the participation of their child in the study
* Absence of opposition of children able to understand the study

Non inclusion Criteria:

* Sickle cell children under the age of 7 or over 17
* Children with mental deficits
* Non-French-speaking parents
* Children receiving only one physiotherapy session and being hospitalized within 24 hours

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: sickle cell children admitted to the paediatric department at the CHR of Orléans
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-04-06 (Actual)

PRIMARY OUTCOMES:
Number of day staying in the pediatric ward according to the maximal inspiratory capacities during incentive spirometry sessions. | throught study completion, an overage of 24hours

SECONDARY OUTCOMES:
Correlation between pain level and maximal inspiratory capacity during incentive spirometry sessions. | throught study completion, an overage of 24hours
Correlation between the maximum inspiratory volume achieved during incentive spirometry and children's mobility (attitude and mobility items according to the EVENDOL scale). | throught study completion, an overage of 24hours
Correlation between the use of analgesic strategies and the inspiratory volume related to patients' size and age | throught study completion, an overage of 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Sandrine PELLETIER, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orleans, Orléans, France

REFERENCES:
- [Result] Bellet PS, Kalinyak KA, Shukla R, Gelfand MJ, Rucknagel DL. Incentive spirometry to prevent acute pulmonary complications in sickle cell diseases. N Engl J Med. 1995 Sep 14;333(11):699-703. doi: 10.1056/NEJM199509143331104. PMID 7637747
- See also: French guidelines for the management of adult sickle cell disease: 2015 update — http://linkinghub.elsevier.com/retrieve/pii/S0248866315600029